CLINICAL TRIAL: NCT03497949
Title: Peri-operative Vasopressor Support in Patients Operated for an Acute Hip Fracture (AHF)
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Bengt Nellgard, Clinical professor, Sahlgrenska University Hospital
Other Study IDs: Hip vasopressor
Record Dates: First submitted 2018-04-10; First posted 2018-04-13 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Hip Fractures; Intraoperative Hypotension
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence of hypotension perioperatively during operation of an acute hip fracture is unknown. As a surrogate factor the usage of vasopressor support is more adequate as the registration of vasopressor drugs are many times not complete in records. The investigators retrospectively investigated the anesthetic journals of 1100 patients with an acute hip fracture (AHF) noting confounding factors and the usage of vasopressors either by injections or infusions and then correlated these results to mortality at 30-, 90- and 365- days

DETAILED DESCRIPTION:
The incidence of hypotension perioperatively during operation of an acute hip fracture is unknown. As a surrogate factor the usage of vasopressor support is more adequate as the registration of vasopressor drugs are many times not complete in records. The investigators retrospectively investigated the anesthetic journals of 1100 patients with an acute hip fracture (AHF) noting confounding factors and the usage of vasopressors either by injections or infusions and then correlated these results to mortality at 30-, 90- and 365-days Confounding factors were; all comorbitity, age, ASA grade as well as type of anesthesia

ELIGIBILITY:
Inclusion Criteria

* Patients with an acute hip fracture

Exclusion Criteria

* Only one fracture within time-limit.
* Unretreivable mortality data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Single center study of patients operated with an acute hip fracture
Sampling Method: Probability Sample
Enrollment: 997 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 365 days

CONTACTS AND LOCATIONS:
Locations (1):
- SahlgrenskaUH, Mölndal, VGR, Sweden